CLINICAL TRIAL: NCT06447870
Title: Research on the Mechanisms of Treatment Non-response in Inflammatory Bowel Disease Based on Multi-omics Technology
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-128
Record Dates: First submitted 2024-05-19; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- primary non-response group: biologic therapy(eg:IFX,ADA,UST,VDZ)
  Interventions: Drug: biologic therapy(eg:IFX,ADA,UST,VDZ)
- response group: biologic therapy(eg:IFX,ADA,UST,VDZ)
  Interventions: Drug: biologic therapy(eg:IFX,ADA,UST,VDZ)

INTERVENTIONS:
Drug: biologic therapy(eg:IFX,ADA,UST,VDZ) — The patients received biologic therapy during the baseline period, and the specific type of medication was determined based on the professional doctor's diagnosis and treatment opinions. Patients were then divided into two groups based on whether primary non-response occurred or not.

SUMMARY:
In recent years, biologic agents such as infliximab, vedolizumab, and ustekinumab have demonstrated tremendous potential in the treatment of inflammatory bowel disease (IBD), altering the traditional treatment paradigm for IBD. Despite their significant efficacy, there remains a subset of patients who do not respond to biologic agents, necessitating research into the response mechanisms of biologic therapy to explore more precise treatment strategies. Preliminary work by the principal investigator has identified multiple potential responder cell subtypes to biologic agents, which may be influenced by the gut and oral microbiota. Therefore, this project proposes to investigate the mechanisms of response to biologic agents, aiming to explore more precise treatment strategies, through the integration of single-cell transcriptomics, 16S rRNA, and other multi-omics technologies on tissue samples, feces, saliva, peripheral blood, etc., from IBD patients before and after treatment. This will involve integrating bioinformatics analysis and in vitro/in vivo functional validation to elucidate the roles of treatment-responsive cell subtypes and gut and oral microbiota in the inflammatory microenvironment of the intestine, with the aim of uncovering the mechanisms of biologic agent therapy and providing new clues for the development of next-generation drug targets.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older; diagnosed with inflammatory bowel disease according to the 2019 European ECCO-ESGAR guidelines; who have not previously received any biologic therapy or, based on the treating physician's judgment, require treatment with infliximab (IFX), adalimumab (ADA), vedolizumab (VDZ), or ustekinumab (UST) after 3 months of medication.

Exclusion Criteria:

* Patients who refuse treatment with infliximab, adalimumab, vedolizumab, or ustekinumab for various reasons, or those with contraindications; patients currently using antibiotics or who have been in contact with probiotics/antibiotics in the past month; those with concomitant active autoimmune diseases, active tumors, etc.; those with severe oral diseases; patients experiencing other diseases unrelated to inflammatory bowel disease during treatment but may affect the efficacy of inflammatory bowel disease treatment; pregnant or lactating women; those deemed unsuitable for participation in this study by the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: based on the treating physician's judgment, The patients require biologic therapy with infliximab (IFX), adalimumab (ADA), vedolizumab (VDZ), or ustekinumab (UST) after 3 months of medication. Patients were then divided into two groups based on whether primary non-response occurred or not.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
clinical response rate | 3 months after biologic therapy began
  The ratio of patients achieving clinical response to the total number of treated patients.
clinical remission rate | 3 months after biologic therapy began
  The ratio of patients achieving clinical remission to the total number of treated patients.

CONTACTS AND LOCATIONS:
Locations (1):
- NanFang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided